CLINICAL TRIAL: NCT06003517
Title: Retrospective Study on Perioperative Safety and Quality Control Based on Real World Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K3120
Record Dates: First submitted 2023-08-13; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Perioperative Complication
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with perioperative safety events: Patients with perioperative safety events, including post extubation tracheal intubation, intraoperative cardiac arrest, allergic reactions.
  Interventions: Procedure: Screening with PSI check list
- Patients without perioperative safety events: Patients without perioperative safety events, including post extubation tracheal intubation, intraoperative cardiac arrest, allergic reactions.
  Interventions: Procedure: Screening with PSI check list

INTERVENTIONS:
Procedure: Screening with PSI check list — Screening PSI with institutional check list

SUMMARY:
Based on the data from the anesthesia record electronic system, patient safety incident (PSI) electronic reporting system and related PSI retrospective cohort in the past 10 years, this project intends to carry out structured and consistent (real world data)RWD processing, and conduct (real world evidence)RWE research related to perioperative safety and quality control in order to characterize the epidemiology of perioperative PSIs, explore the related factors, and construct a prediction model, and on the basis of which to construct a standardized platform for reporting and analysis of perioperative PSIs based on RWD. On this basis, a standardized platform for PSI reporting and analysis was constructed based on RWD.

ELIGIBILITY:
Inclusion Criteria:

* perioperative patients with anesthesia electronic records.
* aged more than 18 years old.

Exclusion Criteria:

* data incomplete
* data missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perioperative patients with anesthesia electronic records that can analysis the patient safety incident.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of PSI | Perioperative period, from the beginning of the surgery to 7 days after the surgery.
  Occurrence of patient safety incident, including post extubation tracheal intubation, intraoperative cardiac arrest, allergic reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided